CLINICAL TRIAL: NCT07066527
Title: Efficacy and Safety Analysis of More Stable Foam and Ordinary Foam Based on Polylauricol in the Treatment of Head and Neck Venous Malformations: a Prospective, Randomized and Controlled Study
Brief Title: Efficacy and Safety Analysis of Polylauric Alcohol More Stable Foam Versus Ordinary Foam in the Treatment of Head and Neck Venous Malformations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202207-006-2
Record Dates: First submitted 2025-03-20; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Venous Malformation
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A common foam prepared from poly (cinnamyl alcohol) (No Intervention): 1% POL solution 2ml + 8ml air was used to produce foam by Tessari's method for head and neck VMs
- More stable foams made from poly -LRB-cinnamyl alcohol) (Active Comparator): 0.05% 0.1 ml hyaluronic acid+1% POL solution 2ml + 8ml air was used to produce foam by Tessari's method for head and neck VMs
  Interventions: Combination Product: The addition of sodium hyaluronate to poly (cinnamyl alcohol-RRB- produces a more stable foam

INTERVENTIONS:
Combination Product: The addition of sodium hyaluronate to poly (cinnamyl alcohol-RRB- produces a more stable foam — According to the study, the half-life of 1% poly (cinnamyl alcohol-RPol(POL) foam with a liquid-to-gas ratio of 1:4 was 142.8(64.32) seconds, in this study, the half-life of the foam made from 1% POL containing 0.05% hyaluronic acid (HA) was 390.4(613.06) seconds, human blood contains a certain amount of HA, according to the literature reported that 0.05% concentration of HA injected into human blood is safe, so this more stable foam preparation method was patented, and published in international journals.
  Arms: More stable foams made from poly -LRB-cinnamyl alcohol)

SUMMARY:
The aim of this study is to explore the efficacy and safety of poly -LRB-cinnamyl alcohol) foam in the treatment of venous malformations of head and neck through a prospective randomized clinical trial, this trial may provide better treatment options and evidence for head and neck VMs.

DETAILED DESCRIPTION:
Foam sclerotherapy is an effective method for the treatment of venous malformations in head and neck, which has been widely used in the world in recent years. The foam hardener is a kind of uniform microfoam formed by the mixture of surfactant liquid hardener and a certain proportion of gas. The microfoam has fluidity and can be injected into the cavity of venous malformation, the foam can replace the blood in the Lacuna, and can expel the blood, the foam occupies the lesion lacuna, makes the hardener be diluted by the blood to the minimum degree, so that the function concentration of the hardener can be guaranteed, the foam can contact the endothelial cells of venous malformations, acting as the contact betthe investigatorsen the liquid hardener and the endothelial cells, and the foam is less mobile than the liquid hardener, so the foam can be replaced by the blood for a longer time than the liquid hardener, sclerosants can affect endothelial cells for a long time. The disadvantage of liquid hardeners is that they are diluted by blood, leading to an insufficient level of desired effect at the injection site and into the normal venous system. In contrast, foam hardeners replace blood rather than mix with it and occupy the interior of blood vessels. The foam blocks blood flow, increasing the time of contact betthe investigatorsen the Hardener and the vessel wall. Foam hardeners are more effective than liquid hardeners in treating VMS. There are many factors that affect the therapeutic effect of foam hardening, such as the types of hardeners and the stability of foam, among which the stability of foam is one of the key factors that affect the therapeutic effect of foam hardening, the stability of the foam is affected by many factors, such as the type, concentration, liquid-gas ratio, gas type and temperature of the Hardener. The half-life, the time it takes for a foam to reduce its volume to half its original volume (half-volume) , is widely used to assess foam stability. According to the study, the half-life of 1% poly (cinnamyl alcohol-RPol(POL) foam with a liquid-to-gas ratio of 1:4 was 142.8(64.32) seconds, in this study, the half-life of the foam made from 1% POL containing 0.05% hyaluronic acid (HA) was 390.4(613.06) seconds, human blood contains a certain amount of HA, according to the literature reported that 0.05% concentration of HA injected into human blood is safe, so this more stable foam preparation method was patented, and published in international journals. Our team used more stable POL foam to treat head and neck VMs, which was found to be safe and effective by retrospective study. The results of this study have been published in international journal. It has also been reported that glycerol added to the sclerosing agent polydocanol or sodium tetradecyl sulfate can enhance the stability of the foam. The foam produced by glycerol has been used in the treatment of VMS of the head and neck for more than 2 years, and that a more stable bubble might work better. Therefore, whether the more stable hardening agent foam will have better therapeutic effect and whether its safety is different from that of ordinary foam, there is only conjecture and no clear evidence to ansthe investigatorsr this question. Therefore, on the basis of the previous research, a prospective randomized clinical trial was conducted to evaluate the efficacy and safety of polycinol foam in the treatment of venous malformations in the head and neck region, this trial may provide better treatment options and evidence for head and neck VMs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-60 years of age, sex unlimited (except pregnant women or those preparing for pregnancy)
2. Clinical diagnosis and imaging () were consistent with head and neck venous malformations
3. Participants volunteered to participate in the trial and signed an informed consent form.

Exclusion Criteria:

1. People with serious systemic diseases, including heart disease, high blood pressure, diabetes, etc. , that are not under control. Heart Attack: 1. Recent frequent attacks of angina. 2. Recent history of myocardial infarction 3. Cardiac function grade iii-iv or with symptoms of sitting breathing, cyanosis, jugular venous distension, lower limb edema, etc. . 4. Heart disease complicated with hypertension 5. Type II or III Type II atrioventricular block, double bundle branch block, as syndrome, diabetes: blood sugar control in 8.88 mmol/L above, hypertension: after taking medicine blood pressure can not be controlled in the normal range namely systolic pressure below 140 mmhg, diastolic pressure below 90 mmhg)
2. Patients who are unable to follow up on time;
3. Persons who are mentally ill or have mental disorders;
4. The patient or his/her authorized person is unwilling to sign a written informed consent or comply with the protocol

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Remission rate of venous malformations in head and neck | 3-4 weeks after treatment
  Patients were satisfied and no further treatment was needed after clinical evaluation. This was the last treatment. The proportion of patients who responded to treatment was counted and compared between the two groups.

SECONDARY OUTCOMES:
Volume of venous malformation | 3-4 weeks after treatment
  The volume changes of venous malformations were compared before and after treatment. The patients were examined by MRI before operation and after the last treatment
Foam injection | 3-4 weeks after treatment
  The total foam volume from the first treatment to the end of treatment was recorded.
Number of treatment | According to the condition whether need to be treated again, is generally 3-4 weeks for a treatment.
  Statistics of patients with the first treatment to the last treatment of the total number of treatments.

CONTACTS AND LOCATIONS:
Overall Officials: shaohua liu, Doctoral, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Shandong University Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No